CLINICAL TRIAL: NCT02143102
Title: vascuCAP: Non-invasive Computer-Aided Phenotyping of Vasculopathy
Brief Title: Non-invasive Computer-Aided Phenotyping of Vasculopathy
Acronym: Q-CAMP
Status: Completed | Type: Observational
Sponsor: Elucid Bioimaging Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 305
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Carotid Atherosclerosis; Peripheral Arterial Disease
MeSH Terms: conditions — Carotid Artery Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After endarterectomy during surgery, the excised plaque specimens will be sent to the hospital's pathology lab to be analyzed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Training set: Data from subjects in the training set will be utilized to further develop the vascuCAPTM classifiers.
- Testing set: Data from subjects in the testing set will be used to assess the study endpoints.

SUMMARY:
The investigators use MRI and/or CT to evaluate the extent, as well as, the structure, composition, and functional aspects of atherosclerotic plaques in human carotid and femoral arteries in patients scheduled to undergo an endarterectomy of the aforementioned vascular beds as part of their routine clinical care.

DETAILED DESCRIPTION:
The investigators hypothesize that in vivo MRI and/or CT examinations of patients, when suitably acquired and analyzed with the vascuCAP™ analysis software, can provide a sufficiently accurate profile of plaque characteristics to provide an objective basis for patient management. Study subjects include patients undergoing endarterectomies to mitigate their clinical risk or symptoms for conditions including stroke, claudication, and critical limb ischemia. The endarterectomy specimens removed at surgery will allow a direct comparison between the MRI information obtained prior to the surgery and the histopathological analyses of the arterial specimens. The vascuCAP™ measurements of structural and functional features of the arterial wall will be performed in patients undergoing endarterectomy. Measured results will be compared in a blinded fashion with histology to assess performance of plaque profiling and build a pilot prediction model for risk scoring.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet one of the following inclusion criteria in order to be eligible to participate in the study:

* Case subjects will be patients with documented carotid atherosclerosis, scheduled for magnetic resonance or CT angiography and subsequent elective endarterectomy with 30 days of enrollment in the study
* Case subjects will be patients with peripheral arterial disease (PAD) with clinical symptoms, scheduled for magnetic resonance or CT angiography and indicated endarterectomy of diseased areas of femoral arteries within 30 days of enrollment in the study

Exclusion Criteria:

* Subjects with claustrophobia or inability to tolerate prior MRI studies.
* Subjects with metal implants that are not MRI compatible (LSU detailed checklist to be attached) including: Subjects with any type of bio-implant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.). Subjects with any type of ferromagnetic bio-implant that could potentially be displaced or damaged, such as aneurysm clips, metallic skull plates, etc.
* Subjects with a history of kidney disease or dialysis that are unable to receive intravenous gadolinium contrast material.
* Female subjects. A urine pregnancy test will be required of all female subjects of childbearing potential prior to inclusion in this study. Pregnant or nursing females will be excluded from the study.
* Subjects who cannot adhere to the experimental protocol.
* Subjects allergic to contrast material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals must meet one of the following inclusion criteria in order to be eligible to participate in the study:
  * Case subjects will be patients with documented carotid atherosclerosis, scheduled for magnetic resonance or CT angiography and subsequent elective endarterectomy with 30 days of enrollment in the study
  * Case subjects will be patients with peripheral arterial disease (PAD) with clinical symptoms, scheduled for magnetic resonance or CT angiography and indicated endarterectomy of diseased areas of femoral arteries within 30 days of enrollment in the study
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-07; Primary Completion 2017-03-14 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Buckler, M.S., Study Director — Elucid Biomaging Inc.
Locations (2):
- United States (2):
  - West Jefferson Medical Center, Marrero, Louisiana
  - LSU ILH, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheahan M, Ma X, Paik D, Obuchowski NA, St Pierre S, Newman WP 3rd, Rae G, Perlman ES, Rosol M, Keith JC Jr, Buckler AJ. Atherosclerotic Plaque Tissue: Noninvasive Quantitative Assessment of Characteristics with Software-aided Measurements from Conventional CT Angiography. Radiology. 2018 Feb;286(2):622-631. doi: 10.1148/radiol.2017170127. Epub 2017 Aug 31. PMID 28858564

RESULTS

PARTICIPANT FLOW:
Groups:
- Development Set: Data from subjects in the training set will be utilized to further develop the vascuCAPTM classifiers.
Period: Overall Study
Arm/Group | Development Set | Testing Set
Started | 97 | 28
Completed | 86 | 28
Not Completed | 11 | 0
Not completed — Lost to Follow-up | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Development Set: Data from subjects in the training set will be utilized to further develop the vascuCAP measurements.
- Total: Total of all reporting groups
Arm/Group | Development Set | Testing Set | Total
Number analyzed (Participants) | 86 | 28 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (11) | 66.6 (10.1) | 66.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 17 | 49
  Male | 54 | 11 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 82 | 25 | 107
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Measurement Bias of Calcification Analyzed by vascuCAP™ Non-invasively Relative to Histopathology as Ground Truth.
Description: Performance of measurements was assessed by estimating the bias (the difference between the measurement and histology)
Time Frame: Assessed on tissue samples collected within 30 days of non-invasive imaging
Measure: Mean (95% Confidence Interval); unit: mm2
Groups:
- Full: Pooled results for final estimation
Arm/Group | Testing Set | Full
Number analyzed (Participants) | 28 | 114
mm2 | -0.47 [-1.75 to 0.41] | .07 [-.22 to .42]

2. Primary Outcome: Measurement Bias of Lipid-rich Necrotic Core Analyzed by vascuCAP™ Non-invasively Relative to Histopathology as Ground Truth.
Description: Performance of measurements was assessed by estimating the bias (the difference between the measurement and histology)
Time Frame: Assessed on tissue samples collected within 30 days of non-invasive imaging
Measure: Mean (95% Confidence Interval); unit: mm2
Arm/Group | Testing Set | Full
Number analyzed (Participants) | 28 | 114
mm2 | 1.26 [.12 to 2.51] | .87 [-.18 to 1.9]

ADVERSE EVENTS:
Time Frame: from time of enrollment through endarterectomy procedure, an average of 1 month
Description: The study protocol was written to ensure that the study have no effect on either diagnosis or treatment of enrollees.
Arm/Group | Development Set | Testing Set
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/28
Other Adverse Events (participants affected / at risk) | 0/86 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-03-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02143102/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT02143102/ICF_001.pdf